CLINICAL TRIAL: NCT01773343
Title: Treatment of Atrophic Acne Scars With a Fractional CO2 Laser at 1 Versus 3 Months Intervals. A Randomized Controlled Trial With Blinded Response Evaluations
Brief Title: Treatment of Atrophic Acne Scars With a Fractional CO2 Laser at 1 Versus 3 Months Intervals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100169; 20110102 (Registry Identifier: 20110102)
Record Dates: First submitted 2013-01-02; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Atrophic Acne Scars
Keywords: skin texture, efficacy, adverse effects
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO2 laser at 1 month interval (Active Comparator): CO2 laser treatment of mild to severe acne scars at 1 month interval
  Interventions: Procedure: Laser
- CO2 laser at 3 monrths interval (Active Comparator): CO2 laser treatment of mild to severe acne scars at 3 month intervals
  Interventions: Procedure: Laser

INTERVENTIONS:
Procedure: Laser — Fractionel CO2 laser: 1 versus 3 months intervals
  Other Names: Fractionel CO2 laser

SUMMARY:
To compare efficacy and adverse effects of fractional CO2 laser of acne scars treatment with 1 versus 3 months intervals

DETAILED DESCRIPTION:
Change in scar texture evaluated by blinded evalutaions. Appearance of erythema, oedema, pigmentation, infection after treatment

ELIGIBILITY:
Inclusion Criteria:

* Have Fitzpatrick skin type I-III. (•Are male or female.
* Are between 18 and 60 years of age.
* Mild to severe acne scarring.
* Are able to read, understand, and sign the Informed Consent.
* Are willing and able to comply with all follow-up requirements -

Exclusion Criteria:

* Have had active localized or systemic infections within 6 months of enrollment
* Have compromised ability for wound healing, such as: malnutrition, oral steroid use, history of collagen vascular disease (e.g. lupus, scleroderma, history of keloid formation (raised and thickened scars), atrophic dermatitis (extreme skin irritation or itchiness) or immunologic abnormalities such as vitiligo (white patches of skin due to loss of pigment)
* Have been treated with lasers, chemical procedures, or other cosmetic procedures on the area to be treated within 6 months of enrollment
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Change in scar texture | 24 weeks

SECONDARY OUTCOMES:
Appearance of erythema, oedema, pigmentation, infection | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lene Hedelund, MD, PhD, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus C, Denmark